CLINICAL TRIAL: NCT00642044
Title: Corneal Collagen Crosslinking With Riboflavin for Keratoconus Treatment: A Brazilian Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Adalmir Morterá Dantas / Department of Ophthalmology Chief, UFRJ - Department of Ophthalmology
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 005/07-CEP
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-03

CONDITIONS: Keratoconus
Keywords: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): The eye with the worst visual acuity receives the treatment. (the other eye serve as control).
  Interventions: Procedure: Corneal Collagen Crosslinking
- B (No Intervention): The eye with the best visual acuity do not receive the treatment.

INTERVENTIONS:
Procedure: Corneal Collagen Crosslinking — UV light and Riboflavin eyedrops every 5 minutes for 30 minutes.
  Arms: A

SUMMARY:
Cross-linking of the cornea increases the mechanical and biochemical stability of the stromal tissue. The purpose of this study is to assess the effectiveness of riboflavin-ultraviolet light induced cross-linking of corneal collagen in improving visual acuity and reducing progression of keratoconus in the Brazilian population.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 35 years.
* Diagnosis of Keratoconus.
* Progression of Ametropia.
* Written informed consent.

Exclusion Criteria:

* Corneal Thickness < 395 micra at thinnest point.
* Other active ocular disease than keratectasia.
* Cornea Guttata.
* Previous ocular surgery.
* Pregnancy.
* Known sensitivity to riboflavin.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Keratometry | 3 months
BSCVA (Best spectacle corrected visual acuity) | 3 months

SECONDARY OUTCOMES:
Endothelial cell count | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Lamy, MD, Principal Investigator — UFRJ
Locations (1):
- Clementino Fraga Filho University Hospital, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Background] Spoerl E, Huhle M, Seiler T. Induction of cross-links in corneal tissue. Exp Eye Res. 1998 Jan;66(1):97-103. doi: 10.1006/exer.1997.0410. PMID 9533835
- [Background] Kolozsvari L, Nogradi A, Hopp B, Bor Z. UV absorbance of the human cornea in the 240- to 400-nm range. Invest Ophthalmol Vis Sci. 2002 Jul;43(7):2165-8. PMID 12091412
- [Background] Sekundo W, Stevens JD. Surgical treatment of keratoconus at the turn of the 20th century. J Refract Surg. 2001 Jan-Feb;17(1):69-73. doi: 10.3928/1081-597X-20010101-09. PMID 11201780
- [Background] Caporossi A, Baiocchi S, Mazzotta C, Traversi C, Caporossi T. Parasurgical therapy for keratoconus by riboflavin-ultraviolet type A rays induced cross-linking of corneal collagen: preliminary refractive results in an Italian study. J Cataract Refract Surg. 2006 May;32(5):837-45. doi: 10.1016/j.jcrs.2006.01.091. PMID 16765803
- [Background] Spoerl E, Mrochen M, Sliney D, Trokel S, Seiler T. Safety of UVA-riboflavin cross-linking of the cornea. Cornea. 2007 May;26(4):385-9. doi: 10.1097/ICO.0b013e3180334f78. PMID 17457183
- [Background] Wollensak G, Spoerl E, Seiler T. Stress-strain measurements of human and porcine corneas after riboflavin-ultraviolet-A-induced cross-linking. J Cataract Refract Surg. 2003 Sep;29(9):1780-5. doi: 10.1016/s0886-3350(03)00407-3. PMID 14522301
- See also: Clementino Fraga Filho University Hospital — http://www.hucff.ufrj.br